CLINICAL TRIAL: NCT02799030
Title: A Randomized Placebo-controlled Clinical Trial of Topical Photodynamic Therapy With 5-aminolevulinic Acid for the Treatment of Actinic Keratosis
Brief Title: A Clinical Trial of Topical Photodynamic Therapy With 5-aminolevulinic Acid for the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biofrontera Bioscience GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALA-AK-CT001
Record Dates: First submitted 2016-05-26; First posted 2016-06-14 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-06

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- BF-200 ALA 0% (Placebo Comparator): Topical application of matched placebo gel without containing 5-ALA. Application of a 1 mm thick layer covering each lesion and approximately 1 cm of the surrounding margin.
  Interventions: Drug: BF-200 ALA 1%; Drug: BF-200 ALA 3%; Drug: BF-200 ALA 10%
- BF-200 ALA 1% (Experimental): Topical application of BF-200 ALA gel containing 0.78 mg/g 5-aminolevulinic acid. Application of a 1 mm thick layer covering each lesion and approximately 1 cm of the surrounding margin.
  Interventions: Drug: BF-200 ALA 1%
- BF-200 ALA 3% (Experimental): Topical application of BF-200 ALA gel containing 3.8 mg/g 5-aminolevulinic acid. Application of a 1 mm thick layer covering each lesion and approximately 1 cm of the surrounding margin.
  Interventions: Drug: BF-200 ALA 3%
- BF-200 ALA 10% (Experimental): Topical application of BF-200 ALA gel containing 78 mg/g 5-aminolevulinic acid. Application of a 1 mm thick layer covering each lesion and approximately 1 cm of the surrounding margin.
  Interventions: Drug: BF-200 ALA 10%

INTERVENTIONS:
Drug: BF-200 ALA 1% — topical treatment for photodynamic therapy combining drug application and after 3 h of drug incubation subsequent illumination with a broad spectrum light source .
  Arms: BF-200 ALA 0%; BF-200 ALA 1%
Drug: BF-200 ALA 3% — topical treatment for photodynamic therapy combining drug application and after 3 h of drug incubation subsequent illumination with a broad spectrum light source .
  Arms: BF-200 ALA 0%; BF-200 ALA 3%
Drug: BF-200 ALA 10% — topical treatment for photodynamic therapy combining drug application and after 3 h of drug incubation subsequent illumination with a broad spectrum light source .
  Other Names: Ameluz
  Arms: BF-200 ALA 0%; BF-200 ALA 10%

SUMMARY:
This was a placebo controlled, double blind, randomized phase II dose-response study to evaluate the efficacy and safety of BF-200 ALA (containing the active ingredient 5 - aminolevulinic acid- ALA) used with photodynamic therapy (PDT) in patients with actinic keratosis (AK).

DETAILED DESCRIPTION:
The study was performed to define the effective therapeutic dose of the active pharmaceutical ingredient (ALA) in a nanoemulsion formulation in the treatment of actinic keratosis (AK) with topical PDT and to assess the efficacy of topical PDT with a new nanoemulsion formulation of ALA in the treatment of AK. The efficacy of BF-200 ALA was calculated by the AK clearance rate, defined as the proportion of AK lesions showing complete remission 12 weeks after PDT treatment.

Subjects of two study centres provided plasma and urine samples for the quantification of ALA and its metabolite, the active photosensitizer protoporphyrin IX (PpIX).

ELIGIBILITY:
Inclusion Criteria:

* The subjects were willing and able to sign the informed consent form.
* Men and women aged between 18 and 85 years.
* Had a general good and stable health condition as confirmed by a physical examination and by medical history.
* The subjects accepted to abstain from sunbathing and the solarium during the study.
* The subjects had at least 3 but not more than 10 clinically confirmed AK target lesion of mild to moderate intensity within the face or bald scalp (excluding eyelids, lips and mucosa), i.e. AK grade I and II. Grade I AK lesions presented as flat, pink maculae without signs of hyperkeratosis and erythema.
* The AK lesions had to be discrete and quantifiable; the distance from one lesion to its neighbour lesion was greater than 1.5 cm.
* The diameter of each AK lesion was not less than 0.5 cm and not greater than 1.5 cm.
* The subjects were free of any significant physical abnormalities (e.g., tattoos, dermatoses) in the potential treatment area that could cause difficulty with examination or final evaluation.
* The subjects were willing to stop using moisturizers and any other topical treatments with anti-aging products, vitamin A, vitamin C, and/or vitamin E containing ointments and creams, and green tea preparations during the study within the treatment area. Sunscreens was allowed, but was not to be applied in the treatment area within approximately 24 hours of a clinic visit with lesion count.
* Only women of childbearing potential who used a highly effective method of contraception and who had a negative serum pregnancy test were allowed to participate in this study.

Exclusion Criteria:

* Had a known hypersensitivity to ALA.
* Had received any other medication known to affect AK 3 months before or during the study.
* Were under immunosuppressive therapy.
* Suffered from porphyria.
* Showed hypersensitivity to porphyrins.
* Suffered from photodermatoses.
* Had inherited or acquired coagulation defects.
* Received medication with hypericin or systemically acting drugs with phototoxic or photoallergic potential within 8 weeks prior to treatment with study drug and PDT
* Had evidence of clinically significant, unstable medical conditions such as

  * a metastatic tumour or a tumour with a high probability of metastatic spread
  * cardiovascular (NYHA class III, IV)
  * immunosuppressive
  * haematological, hepatic, renal, neurological, endocrine
  * collagen-vascular
  * gastrointestinal.
* Subjects with clinically stable medical conditions including, but not limited to the following diseases were allowed to be included into the study, if the medication taken for the treatment of the disease did not match the criteria of the excluded or disallowed medications listed in points 11 and 12 below:

  * controlled hypertension
  * diabetes mellitus type II
  * hypercholesterinaemia
  * osteoarthritis
* Had currently other malignant or benign tumours of the skin within the treatment area (e.g., malignant melanoma, basal cell carcinoma, squamous cell carcinoma).
* Had received the following treatments for any indication in the treatment area within the designated time period before PDT treatment with ALA:
* Topical steroids - 4 weeks
* Topical retinoids - 6 weeks
* Topical diclofenac preparations - 6 weeks
* Topical 5-fluorouracil preparations - 6 weeks
* Topical immunomodulators - 6 weeks
* Surgical excision (except biopsy for diagnostic confirmation) - 6 weeks
* Curettage - 4 weeks
* Cryo-, thermo- or chemodestruction - 6 weeks
* PDT - 6 weeks
* Therapeutic UV-Radiation - 6 weeks
* Had received the following systemic treatments within the designated period before PDT treatment with ALA:
* Interferon - 6 weeks
* Immunomodulators or immunosuppressive therapies - 10 weeks
* Cytotoxic drugs - 6 months
* Investigational drugs - 8 weeks
* Drugs known to have major organ toxicity - 8 weeks
* Corticosteroids (oral or injectable) - 6 weeks
* Inhaled corticosteroids (>1200 µg/day for beclomethasone, or >600 µg/day for fluticasone) - 4 weeks
* A previous treatment with ALA.
* Known allergy to polysorbate 80, caprylic/capric acid triglycerides, isopropyl alcohol, disodium phosphate dihydrate, sodium hydroxide, hydrochloric acid, propylene glycol, methyl parahydroxybenzoate, or propyl parahydroxybenzoate.
* Were known to be pregnant or lactating (currently or within the past 3 months).
* Had any dermatological disease in the treatment area or surrounding area that might be exacerbated by treatment with topical ALA or cause difficulty with examination (e.g. psoriasis, eczema).
* Show cornu cutaneum like alterations of the skin in the face or on the bald scalp (target area).
* Were currently or within the past 8 weeks participating in another clinical study.
* Had active chemical dependency or alcoholism as assessed by the investigator.

  * Topical steroids for the treatment of dermatological diseases (e.g. atopic dermatitis, lichen planus) in locations other than in treatment area were allowed during the study provided the amount used did not exceed 2 mg fluorinated steroids daily for more than 1 week or 6 mg beclomethasone for more than 1 week.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2006-10; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Total clearance rate of AK lesions | 12 weeks after photodynamic therapy (PDT)
  Total clearance rate of all AK lesions, defined as the percentage of baseline lesions within the target treatment areas showing complete remission at week 12 post treatment.

SECONDARY OUTCOMES:
Percentage of subjects totally cleared | 12 weeks after PDT
  Percentage of subject totally cleared, i.e. with complete clearance of all lesions treated 12 weeks after PDT.
Reduction of Total Lesion Area | 12 weeks after PDT
  The reduction of AK lesion area per patient assessed by comparing the total lesion area pre-treatment (at baseline before PDT) and 12 weeks post-treatment
Reduction of Lesion Size | 12 weeks after PDT
  The reduction of the total AK lesion size results from the sum of all single lesion areas by comparing the total lesion size pre-treatment (at baseline before PDT) and 12 weeks post-treatment.
Overall Cosmetic Outcome | 12 weeks after PDT
  Overall Cosmetic Outcome 12 weeks after PDT. The cosmetic outcome at the end-of-study visit will be calculated on the basis of the skin quality assessment (skin surface, hyperpigmentation, hypopigmentation, mottled or irregular pigmentation, degree of scarring, and atrophy. The cosmetic outcome is rated as very good if the sum score of the previously mentioned ratings (all ratings for each sign added up) at a given visit has improved by at least 2 points as compared to baseline; the cosmetic outcome is rated as good if the sum score at a given visit has improved by at least 1 point as compared to baseline; the cosmetic outcome is rated as satisfactory if the sum score at a given visit is identical to the one at baseline; the cosmetic outcome is rated as unsatisfactory if the sum score at a given visit has worsened by 1 point compared to baseline, the cosmetic outcome is rated as impaired if the sum score at a given visit has worsened by at least 2 points compared to baseline.
Local Skin Reactions | during anf after PDT [3h - 4 h]
  Local skin reactions in the treatment area as assessed by the investigator during PDT
Local discomfort | during and after PDT [3h - 4 h]
  Local discomfort or pain reported by the patient during PDT
related Adverse Events (AEs) | up to 12 weeks after PDT
  Frequency and extent of related treatment-emerged AEs (TEAEs ) including related serious AEs

CONTACTS AND LOCATIONS:
Overall Officials: Rolf-Markus Szeimies, Prof Dr, Principal Investigator — Klinikum der Universität Regensburg Klinik und Poliklinik für Dermatologie Franz-Josef-Strauß-Allee 11

IPD SHARING:
Plan to Share IPD: No